CLINICAL TRIAL: NCT04720040
Title: Using YMS-201B in Patients With Mild to Moderate Major Depressive Disorder To Evaluate Efficacy and Safety for the Effect of Improving Depressive Symptoms Open, Single-group, Multicenter Confirmatory Clinical Trial
Brief Title: The Efficacy and Safety of tDCS in Patients With Mild to Moderate Major Depressive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ybrain Inc. (Industry)
Collaborators: The Catholic University of Korea (Other); Inje University (Other); Korea University (Other); Seoul National University Bundang Hospital (Other); Hallym University Medical Center (Other); Soonchunhyang University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YB_ST_SIT1902
Record Dates: First submitted 2021-01-18; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- YMS-201B (Experimental): transcranial Direct Current Stimulation (tDCS) application 5 ~7 days a week for 6 weeks (total of 30~42 applications)
  Interventions: Device: Mind STIM

INTERVENTIONS:
Device: Mind STIM — transcranial Direct Current Stimulation (tDCS) 2mA for 30 min; 30 sec of ramp-up and -down; left (anode) and right (cathode) Dorsolateral prefrontal cortex (DLPFC)

SUMMARY:
This study evaluated the effectiveness and safety of improving depressive symptoms by applying tDCS for 6 weeks to patients with mild to moderate depression.

DETAILED DESCRIPTION:
Patients received tDCS for 30 minutes with an intensity of 1.5 to 2 mA. tDCS was applied over the left (anode) and right (cathode) dorsolateral prefrontal cortex (DLPFC) 5~7 times a week and they were evaluated every 2weeks through questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of a major depressive disorder as confirmed by the DSM-V and MINI (without psychotic features)
* Patients with a K-BDI-II score of 14 or more and 28 or less
* In the case of patients who have previously administered antidepressants, antipsychotics, and anticonvulsants for at least 1 week, Patients with sufficient drug treatment periods of at least 5 times the drug half-life.

Exclusion Criteria:

* Patients diagnosed with Axis I disorders other than major depressive disorder
* Patients diagnosed with other depressive disorders besides major depressive disorder
* Patients who have attempted suicide within 6 months of screening
* Patients who are considered to have problems with EEG and DC stimulation electrode attachment due to scalp deformity, inflammatory reaction, or other dermatological problems
* Patients judged to have other reasons for prohibition of use of tDCS medical devices
* Patients currently taking antidepressants

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2019-12-23 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Korean-Beck Depression Inventory-II | At 6 weeks after treatment.
  Average change of K-BDI-II at 6 weeks after treatment compare to the base respectively. This scale contains 21 questions, each answer being scored on a scale value of 0 to 3. Higher total scores indicate more severe depressive symptoms.The lower the total score, the better the symptoms.

SECONDARY OUTCOMES:
Korean-Beck Anxiety Depression Inventory | Weeks 0, 2, 4, and 6
  The BAI contains 21 questions, each answer being scored on a scale value of 0 (not at all) to 3 (severely). Higher total scores indicate more severe anxiety symptoms.
Hamilton Rating Scale for Depression | Weeks 0, 2, 4, and 6
  The HRSD has been criticized for use in clinical practice as it places more emphasis on insomnia than on feelings of hopelessness, self-destructive thoughts, suicidal cognitions and actions. This scale contained 17items and each item is scored on a 3 or 5point scale. The lower the total score, the better the symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- YBrain Inc., Seongnam-si, Gyeonggi-do, South Korea